CLINICAL TRIAL: NCT03787394
Title: Sensory and Hedonic Effects of FAAA-conjugates Added to Food Products
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL67908.081.18
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Sensory Testing
Keywords: taste enhancers

STUDY DESIGN:
Intervention Model Description: A two-step, randomised controlled intervention study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAAA-enriched (Experimental): food products enriched with FAAA-conjugates
  Interventions: Other: adding taste enhancer
- Plain (Placebo Comparator): Food products without FAAA-conjugates
  Interventions: Other: adding taste enhancer

INTERVENTIONS:
Other: adding taste enhancer — Comparing sensory profiles of food products either enriched with FAAA-conjugates or plain

SUMMARY:
Rationale: According to preliminary observations provided by the research and development department (R&D) of Givaudan, addition of specific fatty acid-amino acid (FAAA)-conjugates to a wide range of food products resulted in an enhancement of several sensory and hedonic effects. Such effects could be attributed to the so-called kokumi sensation, a taste concept that has been described as a "taste enhancer" that magnifies and lengthens all the other five basic tastes. The exact mechanisms of the kokumi sensation are as of yet unclear. Perception of the kokumi sensation depends on the context of other taste compounds and integration into food matrices. A systematic investigation is necessary to objectively evaluate whether the addition of specific FAAA-conjugates results in the enhancement of sensory and hedonic effects. Furthermore, we want to assess the dependency of these effects on the food matrix. To do so, a combination of discrimination, descriptive and hedonic testing will be carried out.

Objectives: The primary objectives are: to determine if there is a perceivable difference between plain and FAAA-enriched versions of selected food products and describe sensory and/or hedonic differences between them; to assess the dependency of FAAA-conjugates on the food matrix.

Study design: A two-step, randomised controlled intervention study will be carried out. Study population: 40 healthy, adult (18-55 years) males and females (BMI 18 - 27 kg/m2) from Wageningen and surroundings will be included.

Intervention (if applicable): FAAA-conjugates: in step one, FAAA-conjugates will be integrated into food products; in step two, FAAA-conjugates will both be administered separately (using a tasteless mouthwash) and integrated into food products.

Main study parameters/endpoints: The primary outcome parameters are: proportion of correct answers (discrimination testing); sensory evaluation score means (descriptive testing); and hedonic evaluation score means (hedonic testing).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The current study is non-therapeutic to subjects. Risks associated with participation are negligible and compared to other studies, the burden can be considered low. The FAAA-conjugates used in the intervention are declared "generally recognised as safe" (GRAS) by the Flavour Extract Manufacturers Association (FEMA) and pose no known adverse health effects.

DETAILED DESCRIPTION:
FAAA conjugates are compounds containing different long-chain fatty acids and simple amino acids. They are involved in multiple signalling pathways playing a role in the regulation of homeostatic and non-homeostatic eating behaviour (Jager & Witkamp, 2014). FAAA-conjugates are naturally occurring in various animal and plant food sources, yet their dietary relevance and exact mechanism of action remains unclear. Notwithstanding, they have been related to improved food sensations and hedonic effects (Jager & Witkamp, 2014; Witkamp, 2018; Yoshida et al., 2013). FAAA compounds have been declared GRAS by FEMA, which guarantees their safe use in commercially available food products (Flavour Extract Manufacturers Association, 2018).

According to preliminary observations provided by the research and development department (R&D) of Givaudan, the addition of specific FAAA-conjugates to a range of food products resulted in an enhancement of several sensory- and hedonic effects in product evaluation. Panellists reported accentuated palatability; aftertaste masking; enhanced fat, sweet, salt and umami perception; and mouthfeel improvement. However, the reproducibility of these results is questionable, as substantial variation in the effects arose both within and between a small sample of volunteers. It is unclear whether these effects are specific for and dependent on integration of these conjugates in a certain food matrix, or if they have a more general boosting effect, relevant for taste or flavour. Perhaps the boosting effect also affects other sensory domains (e.g. vision).

The aforementioned reported sensory/hedonic effects could be attributed to what has been described in literature as the kokumi sensation, which is related to activation of calcium-sensing receptors on the human tongue, albeit the exact mechanism remains to be elucidated (Feng, Zhang, Zhuang, Zhou, & Xu, 2016; Kuroda & Miyamura, 2015; Ohsu et al., 2010). Although Kokumi is associated with taste perception, it is most likely not a primary taste, since its effects exist in the context of other taste compounds. On their own, kokumi compounds elicit only very slight or no taste sensations but incorporated in a food matrix they can enhance other taste sensations. The threshold concentration of kokumi compounds in a plain water solution to induce a taste sensation is usually very high, while the threshold concentration in food to enhance other taste sensations can be very low. (Dunkel, Koster, & Hofmann, 2007; Feng et al., 2016; Kuroda & Miyamura, 2015).

On the basis of preliminary testing done by R&D Givaudan, the study described in the current protocol aims to systematically investigate the sensory and hedonic effects of FAAA-conjugates. To do so, specific FAAA-conjugates will be integrated into two food products (one sweet (chocolate milk) and one savoury (salad dressing), which will be sensorially and hedonically evaluated. Furthermore, the dependency of FAAA-conjugates on the food matrix will be studied by administering them separately from food products. An untrained panel will be used, since consumers are not only capable of providing accurate and reliable information about product sensory characteristics, but can also serve as a measure of potential performance of the product in the marketplace (Ares & Varela, 2017; Lawless & Heymann, 2010).

If results are in line with the aforementioned preliminary observations, they can add to the body of knowledge and underpin future studies investigating the kokumi sensation and the mechanistic background of FAAA-conjugate effects. Moreover, food product reformulation with the use of FAAA-conjugates could positively impact a wide range of consumers. Due to their boosting sensory/hedonic effects, enriching foods with FAAA-conjugates has the potential to reduce sugar, fat and salt content in a wide range of food products without compromising on experienced flavour, thereby reducing sugar, fat and salt intake and their harmful effects. More importantly, the elderly and seriously ill patients could benefit from the palatability-enhancing effects ascribed to kokumi molecules, which could stimulate appetite and help reverse weight loss (Witkamp, 2018).

2. OBJECTIVES

Primary Objective(s):

The primary objective of the current study is to determine if there is an objective perceivable difference between plain and FAAA-enriched versions of selected food products and describe sensory and/or hedonic differences between them, using a combination of discrimination testing, descriptive analyses and hedonic tests.

Secondary Objective(s):

The secondary objective is to assess the dependency of FAAA-conjugates on the food matrix, by separating administration of compound and product and assessing how separation affects sensory and hedonic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55 years
* BMI: 18.0 - 27.0 kg/m2
* Healthy (as judged by subject)
* Consumer of products used in the study
* Proficient in spoken and written English.

Exclusion Criteria:

* Failure to meet any of the inclusion criteria
* Weight loss or weight gain of 5 kg or more during the last 2 months
* Regular smoker (> 1 cigarette per day);
* Restrained eater, assessed by the DEBQ (score of >2.37 for men and >3.24 for women (van Strien, Frijters, Bergers, & Defares, 1986))
* Pregnant or lactating woman
* Anosmia or ageusia (self-reported)
* Food allergies or intolerances relevant for the food products used in the experiment
* Student/employee of the WUR Sensory Science and Eating Behaviour department

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-09 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
discrimination test | 90 minutes
  percentage correctly identified FAAA-enriched samples
descriptive tests | 45 minutes
  ratings sensory attributes on VAS-scales
hedonic test | 45 minutes
  ratings product liking on VAS-scales

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Jager, PhD, Principal Investigator — Wageningen University, Division of Human Nutrition

IPD SHARING:
Plan to Share IPD: No